CLINICAL TRIAL: NCT05916560
Title: A Parallel-Group, Single-Dose, Phase 1, Open-Label Study to Investigate the Pharmacokinetics of LY3437943 in Participants With Hepatic Impairment Compared With Healthy Participants
Brief Title: A Study of LY3437943 in Participants With Impaired and Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18531; J1I-MC-GZBT (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Hepatic Insufficiency
Keywords: Pharmacokinetics; Hepatic Impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — retatrutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3437943 (Normal Hepatic Function) (Experimental): LY3437943 administered subcutaneously (SC).
  Interventions: Drug: LY3437943
- LY3437943 (Severe Hepatic Impairment) (Experimental): LY3437943 administered SC.
  Interventions: Drug: LY3437943
- LY3437943 (Moderate Hepatic Impairment) (Experimental): LY3437943 administered SC.
  Interventions: Drug: LY3437943
- LY3437943 (Mild Hepatic Impairment) (Experimental): LY3437943 administered SC.
  Interventions: Drug: LY3437943

INTERVENTIONS:
Drug: LY3437943 — Administered SC.

SUMMARY:
The main purpose of this study is to measure how much of LY3437943 gets into the bloodstream and how long it takes the body to eliminate it in participants with mild, moderate and severe impaired liver function compared to healthy participants with normal liver function. The safety and tolerability of LY3437943 will also be evaluated. The study may last up to 9 weeks for each participant including the screening period.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Have a body mass index within the range 19.0 to 42.0 kilograms per meter squared (kg/m²), inclusive
* Healthy or various degrees of hepatic impairment depending on the study group

Exclusion Criteria:

Participants with hepatic impairment:

* Have or are anticipating an organ transplant within the next 6 months
* Requires needle evacuation of ascites fluid more than 2 times per month
* Have had variceal bleeding within 3 months of check-in, unless the participant has undergone a successful banding procedure; in that case, may check-in from 1 month after the banding procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve from time zero to infinity (AUC0-∞) of LY3437943 | Predose up to 30 days postdose
  PK: AUC0-∞ of LY3437943
PK: Maximum observed concentration (Cmax) of LY3437943 | Predose up to 30 days postdose
  PK: Cmax of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Arizona Clinical Trials - Chandler, Chandler, Arizona
  - Accel Research Sites- Clinical Research Unit, DeLand, Florida
  - Advanced Pharma Clinical Research, Miami, Florida
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No